CLINICAL TRIAL: NCT05397249
Title: The Impact of Mindfulness and Spirituality on Student Well-being-Efficacy Study
Brief Title: The Impact of Mindfulness and Spirituality on Student Well-being
Acronym: MSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Gulden Esat, Doctoral Student, University of Houston
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001119
Record Dates: First submitted 2019-11-11; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Well-being; Stress; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Mindfulness; Spiritual Therapies

STUDY DESIGN:
Intervention Model Description: This study is designed as an experimental longitudinal study using a 2 X 3 factorial repeated measures design. The 2 level factor is mindfulness and mindfulness plus spirituality. The 3 level factor is the dose of the intervention (i.e., control, one class a week, and two classes a week).
Who Masked: Participant
Masking Description: Participants are blind to their conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Mindfulness only training (Experimental): Face to face twice weekly 10 minutes training of Mindfulness only training.
  Interventions: Behavioral: Mindfulness Training
- Mindfulness with spirituality (Experimental): Face to face twice weekly 10 minutes training of Mindfulness only training plus the Spirituality components.
  Interventions: Behavioral: Mindfulness Training
- Low dose Mindfulness only (Experimental): Face to face once weekly 10 minutes training of Mindfulness only training.
  Interventions: Behavioral: Mindfulness Training
- Low dose Mindfulness with Spirituality (Experimental): Face to face once weekly 10 minutes training of Mindfulness only training plus the Spirituality components.
  Interventions: Behavioral: Mindfulness Training
- No treatment (No Intervention): No intervention is being delivered, however, participants are led to believe that they are receiving some degree of a mindfulness training embedded in their regular course curriculum.

INTERVENTIONS:
Behavioral: Mindfulness Training — The participants are given strategies of mindfulness, asked to complete worksheets and participate in meditations.
  Other Names: Mindfulness only or Mindfulness with Spirituality
  Arms: Low dose Mindfulness only; Low dose Mindfulness with Spirituality; Mindfulness only training; Mindfulness with spirituality

SUMMARY:
The purpose of this research is to find effective ways of well-being promotion in higher education settings. A unique mindfulness training was developed that includes cognitive, emotional, social, and spiritual components. The training is being delivered during class-time of the following courses: Personal Development and College Success, Understanding Health Behavior, and Health Promotion and Disease Prevention. The objective of the study is to explore the training in regard to dosage effects and the incremental effect of spirituality. While the proximal targets of the intervention are well-being and stress, the ultimate targets are grades and persistence in college.

The hypotheses to be tested are:

* Mindfulness training will increase the well-being and decrease the stress, anxiety and depression symptomology of the participants.
* Mindfulness training will increase the functioning of the participants measured through GPA and hours spent in community engagement.
* The "mindfulness training with spiritual components" will have a greater impact than the "mindfulness only training" on well-being.

The study is designed as an experimental longitudinal study using a 2 X 3 factorial repeated measures design. The 2 level factor is mindfulness and mindfulness plus spirituality. The 3 level factor is the dose of the intervention (i.e., control, one class a week, and two classes a week).

DETAILED DESCRIPTION:
This study is the efficacy study of the MSW pilot study (#519)(Fall 2017 and Spring 2018). It will have about 200 participants and will use biometric measures such as salivary cortisol and sleep quality, in addition to the self-report measures. The participants are the HDFS 1311 Personal Development and College Success, HLT 3301 Understanding Health Behavior Theory and Practice, and HLT3381 Health Promotion and Disease Prevention courses students. Two sections of the HDFS 1311 course were assigned to Mindfulness only, and Mindfulness with Spirituality training; another two sections are low-dose control groups, and one section is the no-treatment control group. HLT 3301 is assigned to be Mindfulness only, HLT3381is Mindfulness with Spirituality.

Acceptability and feasibility of the mindfulness training were pilot-tested during the 2017-2018 academic year. Participants thought that the training was helpful, engaging, practical, understandable, pleasant, and relevant to their life as a student at a rate between 94- 100%. The study defines spirituality as the diffusion of the transcendental meaning over the relationship with the self, the immediate social environment, and consequently the wider world. Thus, spirituality can potentially create meaning and purpose in one's life, a variable of which predicts academic self-regulation and GPA and positively related to the treatment of depression and anxiety.

The self-report measures are Pemberton Happiness Index; Five Facet Mindfulness Scale; Intrinsic Spirituality Scale; DASS Depression, Anxiety and Stress Scale; and Pittsburg Sleep Quality Index. The participants' GPA will be accessed through the UH Records Office if FERPA conditions are met.

The baseline data were collected at the beginning of the Fall semester and will be collected at the end of the semester. Additional follow-up data will be collected at the end of the Spring semester. The proximal outcomes of the study are well-being, stress, anxiety, depression, and fall semester grades. Adherence to intervention, intervention delivery quality, and participant engagement are going to be controlled through checklists filled by independent observers; instructor effect will be controlled by rotating the instructors.

The groups will be compared on all of the variables involved in this study, examining for dosage effects and effects of spirituality. There will also be an analysis of correlations between variables, such as the correlation between well-being and grades. The group comparison data have a multilevel structure, with repeated measures nested within individuals and individuals nested in classrooms. The initial plan is to conduct a 2X3 repeated measures ANOVA. If there are large differences in the groups on participant characteristics at baseline, a 2 X 3 ANCOVA will be used. If there are large intraclass correlations in the nested data, investigators will conduct multi-level modeling to examine group differences.

ELIGIBILITY:
Inclusion Criteria: College students over 18. -

Exclusion Criteria: None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in GPA | Collected at the beginning of the semester before the intervention started and at the end of the semester within two weeks period (November and December 2018), and 5 months after the completion of the intervention (May 2019)
  Unofficial, and official GPA records collected through permission granted by the participants. UH uses a 4 point GPA scale, higher score representing better academic achievement. The highest and lowest scores are 4 and 0.
Change in reported well-being score measured by Pemberton Happiness Index | Study had 3 iterations. For all, data is collected at the beginning and end of the semester, before the intervention started, and at the end of the intervention. For 1 iteration, follow up data was collected 5 months after the intervention ended.
  Pemberton Happiness Index(PHI) is a self-report measure that measures the degree of agreement to the 11 statements such as "I am very satisfied with my life". A 10-point Likert scale is used, the high score representing better well-being. Also, it has another section that asks for 10 positive and negative events that happened yesterday through a Yes/No checklist. This leads to another score highest 10, lowest 0, which is added to the total score of the previous 11 items. The highest and lowest scores are 120 and 0.
  PHI yields four types of well-being scores: General, hedonic, eudaimonic, social
Change in depression, anxiety, stress symptoms measured by Depression Anxiety Stress Scale | Study had 3 iterations. For all, data is collected at the beginning and end of the semester, before the intervention started, and at the end of the intervention. For 1 iteration, follow up data was collected 5 months after the intervention ended.
  Depression Anxiety Stress Scale (DASS) is a self-report measure that asks the participants about the symptoms of depression, anxiety, and stress as they apply to them in the past week. It uses a 4 point Likert scale, the highest score representing more intense experience of symptoms. The highest and lowest scores are 63 and 0.
salivary cortisol levels measured by Enzyme Immunoassay Technique | At the end of semester (November 2018) collected within a week period.
  Saliva was collected from the two intervention groups and sent to the laboratory for analysis of the cortisol level found.
time spent in deep, light, and REM sleep measured by activity tracker | At the end of semester (November 2018) collected within a week period.
  Sleep quality was tracked with activity trackers from the two intervention groups. Students wore a Fitbit device for three days.
Change in sleep quality measured by Pittsburgh Sleep Quality Index | Collected only for the first iteration of the study:at the beginning and end of the semester, before the intervention started, and at the end of the intervention. For 1 iteration, follow up data was collected 5 months after the intervention ended.
  PSQI- Pittsburgh Sleep Quality Index is a self-report measure that uses a 4 point Likert scale of frequency that represents the problems encountered related to the quality of sleep (Cannot get to sleep within 30 minutes). The higher frequency would yield to a lower sleep quality index score. The highest and lowest scores are 57 and 0.
Change in Community Involvement | Collected only for the first iteration of the study:at the beginning and end of the semester, before the intervention started, and at the end of the intervention. For 1 iteration, follow up data was collected 5 months after the intervention ended.
  Self-report of community involvement through a Yes/No response to the following question: Are you involved in any community service (church, non-profit organization, or individual)?

SECONDARY OUTCOMES:
Change in reported mindfulness score measured by Five Facet Mindfulness Questionnaire | Collected only for the first iteration of the study:at the beginning and end of the semester, before the intervention started, and at the end of the intervention. For 1 iteration, follow up data was collected 5 months after the intervention ended.
  Five Facet Mindfulness Questionnaire is a self-report measure that uses a 5 point Likert scale to represent the opinion of the participants about the presented statements in terms of its intensity . "When I'm walking, I deliberately notice the sensations of my body moving." is an example item that participants mark how true it is for them (never or always true). Highest score represents a higher mindfulness quality. Possible highest and lowest scores are 195 and 39.
Change in reported spirituality measured by Intrinsic Spirituality Scale | Collected only for the first iteration of the study:at the beginning and end of the semester, before the intervention started, and at the end of the intervention. For 1 iteration, follow up data was collected 5 months after the intervention ended.
  The Intrinsic Spirituality Scale is a self-report measure using a degree of agreement scale with 10 Likert points. The items are stated to prompt the participants to choose their level of spirituality. The following is an example item: In terms of the questions I have about life, my spirituality answers no questions ( a score of 0), or all of my questions ( a score of 10). The possible highest and lowest scores are 60 and 0, the highest score indicating a higher spirituality level.
Change in reported affect measured by Positive and Negative Affect Schedule- Calm-Focus | Collected for the second and third iterations of the study at the beginning and and at the end of each mindfulness lesson. The lessons lasted between 10 to 15 minutes.
  The measure assesses positive and negative emotions in children and adults. The measure includes 10 items consisting of single words indicating positive and negative affect (e.g. sad, happy, scared, cheerful). The scale had two more items measuring "calm" and "focus" which are conceptualized to represent a mindfulness state. Participants are asked to rate how often they have felt this way during the past week using a 5-point scale with responses: never, a little, moderately, quite a bit, and extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Gulden H Esat, PhD, Principal Investigator — University of Houston; Bradley H Smith, Study Chair — University of Houston
Locations (2):
- United States (2):
  - University of Houston, Houston, Texas
  - Gulden Esat, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Raw data of self-report data will be shared.
Supporting Information: Study Protocol
Time Frame: August 2020
Access Criteria: Researchers need to contact the PI to request the data.